CLINICAL TRIAL: NCT00086294
Title: 5HT2A/C Serotonin Blockade in Parkinson's Disease
Brief Title: ACP-103 to Treat Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040225; 04-N-0225
Record Dates: First submitted 2004-06-29; First posted 2004-06-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-11-15

CONDITIONS: Parkinson's Disease; Dyskinesias
Keywords: Non-Dopaminergic; Dyskinesias; Fluctuations; Inverse Agonist; ACP-103; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — pimavanserin

INTERVENTIONS:
Drug: Intravenous Levodopa
Drug: ACP-103

SUMMARY:
This study will evaluate the effects of an experimental drug called ACP-103 on Parkinson's disease symptoms and on dyskinesias (involuntary movements) that develop as a result of long-term levodopa treatment. ACP-103 changes the spread of certain brain signals that are affected in patients with Parkinson's disease.

Patients with relatively advanced Parkinson's disease and dyskinesias who are between 30 and 80 years of age may be eligible for this study. Candidates are screened with a complete medical history and physical examination, neurological evaluation, blood and urine tests, and electrocardiogram (ECG). A brain magnetic resonance imaging (MRI) scan, CT scan, and chest x-ray may be done if medically indicated.

Patients enrolled in the study will, if possible, stop taking all antiparkinsonian medications for one month (2 months for Selegiline) before the study begins and throughout its duration. Exceptions are Sinemet (levodopa/carbidopa), Mirapex (pramipexole) and Requip (ropinirole).

Levodopa Dose Finding

After the screening evaluations, patients are admitted to the NIH Clinical Center for 2 to 3 days to undergo a levodopa "dose-finding" procedure. For this test, patients stop taking Sinemet and instead have levodopa infused through a vein. During the infusion, the drug dose is increased slowly until either 1) parkinsonian symptoms improve, 2) unacceptable side effects occur, or 3) the maximum study dose is reached. Side effects are monitored closely during the infusions, and parkinsonian symptoms are evaluated frequently during and after the infusions. The infusions usually begin early in the morning and continue until evening. Once the infusion is finished, patients resume taking their regular oral Sinemet dose. The infusions are repeated once a week during 1-day inpatient evaluations.

Treatment

Patients are randomly assigned to take either ACP-103 followed by placebo (a look-alike pill with no active ingredient) once a week for 10 weeks or vice versa (placebo followed by ACP-103). Patients are admitted to the Clinical Center for each dose. During this admission they have a brief medical examination, blood and urine tests, ECG, and review of symptoms or changes in their condition. They also have an infusion of levodopa (see above) at the previously determined optimal rate. Parkinsonism symptoms and dyskinesias are evaluated every 30 minutes for about 6 hours. At the end of the infusions and ratings, patients are discharged home with their regular Parkinson's medications until the following visit.

Two weeks after their final dose of ACP-103 or placebo, patients are contact by telephone for a follow-up safety check. At that time, the investigator may ask the patient to return to the clinic for closer evaluation.

DETAILED DESCRIPTION:
Introduction: In Parkinson's disease (PD), levodopa-induced dyskinesias and motor fluctuations are frequent, disabling complications. Therefore, it is imperative to find nondopaminergic approaches to the palliation of parkinsonian signs. Previously, we demonstrated that drugs that block 5HT2A receptors benefit motor dysfunction in parkinsonian animals.

Objective: To test our hypothesis that blockade of serotonin 2A/2C receptors (5HT2A/C) will lessen the severity of parkinsonian signs and levodopa-associated motor response complications in PD patients.

Methods: In a placebo-controlled, proof-of-principle study, the effect of the 5HT2A/C receptor inverse agonist ACP-103 on levodopa induced motor complications and parkinsonian signs will be assessed in up to 20 patients with moderately advanced Parkinson's disease. Efficacy will be assessed through the use of validated motor function scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

Risks and benefits: Risks involved in this study are a minor increase over minimal risks and are deemed reasonable in relation to potential benefits. This investigation should lead to a better understanding of the pathophysiology and treatment of levodopa-induced motor complications in PD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who meet all of the following inclusion criteria will be eligible to participate in the study:

1. Patient is between the ages of 30 and 80 (inclusive);
2. Patient has been diagnosed with idiopathic Parkinson's disease based on the presence of a characteristic clinical history and neurological findings;
3. Patient has relatively advanced disease with levodopa-associated motor response complications, including peak-dose dyskinesias and wearing-off fluctuations;
4. Patient is willing to adhere to protocol requirements as evidenced by written, informed consent.

EXCLUSION CRITERIA:

Patients meeting any of the following exclusion criteria will not be enrolled or will be immediately excluded from the study, as appropriate:

1. Patient has a history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk, including bronchospasm or lung disease, renal and hepatic disease, clinically significant cardiac arrhythmias and/or myocardial ischemia;
2. Patients with clinically significant orthostatic hypotension;
3. Patient has clinically significant laboratory abnormalities including renal and hepatic functions elevation greater than twice the upper limit of normal;
4. Patient is unable to be treated with levodopa/carbidopa alone or with a single, relatively short-acting dopamine agonist, such as pramipexole or ropinirole;
5. Patient is taking a prohibited concomitant medication as listed below:

   The following medications are forbidden for at least one month prior to randomization and during the course of the study:
   * Anticoagulants: etomidate, erythromycin, oral azole antifungals, cyclosporine, cisapride, astemizole;
   * NMDA antagonists: e.g. amantadine, budipine, memantine, remacemide, dextromethorphan;
   * Any other investigational drug;
   * Drugs which are not used primarily to treat Parkinson's disease but which may modify parkinsonian symptoms: neuroleptics, metoclopramide, compazine, beta blockers;
   * Drugs with significant muscarinic receptor antagonist activity: Cogentin, Akineton, Artane, Ditropan, Detrol, Elavil, Anafranil, Norpramine, Sinequan, Tofranil, and Pamelor;
   * Drugs known to improve dyskinesias: amantadine, dextromethorphan, beta-blockers, fluoxitene, clozapine, quetiapine, olanzapine, buspirone, other anxiolytics, antipsychotics, cannabinoid receptor antagonists, adenosine A2a antagonist;
   * Drugs known to exacerbate dyskinesias: sodium valproate, CNS stimulants;
   * Drugs known to have 5HT receptor affinity: ritanserin, sumatriptan
   * Drugs known to interact with serotonergic mechanisms excluding 5HT3 receptor based antiemetics;
   * Dopamine agonists known to have a relatively long half-life: cabergoline and pergolide.
6. Patient who has not been using or unwilling to continue using an adequate contraceptive method (such as oral contraception, surgical sterilization, IUD, diaphragm in conjunction with spermicidal foam and condom on the male partner, or systemic contraception) for the last 30 days, or is not at least one year post-menopausal (if female);
7. Patient is pregnant or breastfeeding;
8. Patient has prior bilateral pallidotomy or other ablative surgeries for treatment of PD;
9. Patient has cognitive impairment (MMSE less than 24);
10. Patient has participated in a clinical study with an investigational drug within the last 30 days;
11. Patient has a condition (such as active drug or alcohol abuse) that, in the opinion of the investigators, would interfere with compliance or safety;
12. Patient is unwilling to sign an informed consent or to comply with protocol requirements.
13. Any previous exposure to ACP-103

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-06-25; Study Completion 2007-11-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mizuno Y, Mori H, Kondo T. Parkinson's disease: from etiology to treatment. Intern Med. 1995 Nov;34(11):1045-54. doi: 10.2169/internalmedicine.34.1045. PMID 8774962